CLINICAL TRIAL: NCT03786939
Title: Evaluation of Outcomes of Coronary Artery Bypass Grafting.
Acronym: EOCABG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EOCABG
Record Dates: First submitted 2018-12-20; First posted 2018-12-26 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-10

CONDITIONS: Ischemic Heart Disease; Coronary Artery Bypass Grafting
Keywords: Ischemic Heart Disease; coronary artery bypass grafting; on-pump CABG; off-pump CABG; pump - assisted CABG; myeloperoxidase after CABG
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- On-pump CABG. (Other): On-pump CABG.
  Interventions: Procedure: On-pump CABG.
- Off-pump CABG. (Other): Off-pump CABG.
  Interventions: Procedure: Off-pump CABG.
- Pump-assisted CABG. (Other): Pump-assisted CABG.
  Interventions: Procedure: Pump-assisted CABG.

INTERVENTIONS:
Procedure: On-pump CABG. — On-pump coronary artery bypass grafting.
  Arms: On-pump CABG.
Procedure: Off-pump CABG. — Off-pump coronary artery bypass grafting.
  Arms: Off-pump CABG.
Procedure: Pump-assisted CABG. — Pump-assisted CABG.
  Arms: Pump-assisted CABG.

SUMMARY:
Evaluation of outcomes of coronary artery bypass grafting.

DETAILED DESCRIPTION:
Evaluation of outcomes of coronary artery bypass grafting (CABG) on-, off- pump, pump assisted as well as bimammary coronary artery bypass grafting.

Objective:

To assess myocardial ischemic-reperfusion damage during different kinds of CABG.

To assess complications after during different kinds of CABG.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic heart disease with indications for coronary artery bypass grafting.

Exclusion Criteria:

* valve disease

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-12-20 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Death. | 30 days during in stay.
  Death during in-stay.

SECONDARY OUTCOMES:
Death over 1 year after CABG. | 1 year.
  Death over 1 year after CABG.
Death over 3 year after CABG. | within 3 years.
  Death over 3 year after CABG.
Death over 5 year after CABG. | within 5 years.
  Death over 5 year after CABG.
Acute myocardial infarction after CABG. | within 30 days after CABG
  Acute myocardial infarction (Criteria: troponin I>10+ST-elevation ECG+hemodynamic instability - record in medical history ot Cardiac Index<2.3).
Acute myocardial infarction after CABG. | within 1 year after CABG
  Acute myocardial infarction (Criteria: troponin I>0.05+ST-elevation on ECG).
Acute myocardial infarction after CABG. | within 3 years after CABG
  Acute myocardial infarction (Criteria: troponin I>0.05+ST-elevation on ECG).
Acute myocardial infarction after CABG. | within 5 years after CABG
  Acute myocardial infarction (Criteria: troponin I>0.05+ST-elevation on ECG).
Shunt dysfunction during 30 days after CABG. | within 30 days after CABG
  Criteria: Stenosis or occlusion of graft on coronary angiography.
Shunt dysfunction during 1 year after CABG. | within 1 year after CABG
  Criteria: Stenosis or occlusion of graft on coronary angiography.
Shunt dysfunction during 3 years after CABG. | within 3 years after CABG
  Criteria: Stenosis or occlusion of graft on coronary angiography.
Shunt dysfunction during 5 years after CABG. | within 5 years after CABG
  Criteria: Stenosis or occlusion of graft on coronary angiography.
Stroke. | within 30 days after CABG
  Stroke after CABG (Record of neurologist in medical history or/and MRI findings).
Renal Dysfunction. | within 30 days after CABG
  Increase serum creatinine level greater than 25% of reference value after CABG.
Atrial fibrillation. | within 30 days after CABG
  New onset of atrial fibrillation after CABG (ECG findings: f-waves).
IABP | within 30 days after CABG
  Intra-Aortic Balloon Pump (non - planned intervention aftet CABG due to hemodinamic instability (Cardiac Index <2.3))
Infection or febrile. | within 30 days after CABG
  Infection or febrile (leucocytosis > 9.0 more than 7 days after CABG or CRP > 10 or t>37.0 more than 7 days after CABG).
Residual myocardial ischemia. | within 30 days after CABG
  New onset of myocardial contractility deterioration on echocardiography (with or without strain, documented hypokinetic or akinetic wall motion).

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Nemkov, PhD, Study Director — First State Pavlov Medical University
Locations (1):
- First Pavlov State Medical University, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No
Individual participant data are confidential.